CLINICAL TRIAL: NCT06635668
Title: Baseline ACL Injury Risk Screening and Normative Data
Status: Recruiting | Type: Observational
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Other Study IDs: ACL- BUS
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: ACL Injury; Anterior Cruciate Ligament Injuries; Musculoskeletal Injury
Keywords: Athletes; Biomechanics
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational cohort study aimed at establishing a database of normative biomechanics for healthy athletes and surveying these athletes for one year following baseline testing for the occurrence of new musculoskeletal injuries, with a particular emphasis on ACL injuries.

DETAILED DESCRIPTION:
This study is a prospective, observational cohort study aimed at establishing a database of normative biomechanics data for healthy athletes. The primary focus is on quantifying muscle strength, movement patterns, and biomechanics in relation to the risk of musculoskeletal injuries, particularly ACL injuries. The study will also explore the relationship between these biomechanical factors and the occurrence of new injuries over a one-year follow-up period.

The research will involve a large sample size of athletes within the Sanford Health service area, including those participating in organized sports at middle schools, high schools, and universities. Advanced marker less three-dimensional motion capture technology will be employed to gather high-fidelity biomechanical data. This will allow for the development of sophisticated algorithms to assess individual injury risk and facilitate targeted interventions aimed at reducing the likelihood of ACL injuries.

Participants will undergo an injury risk screen, which is a standard component of the athletic camps sponsored by Sanford Sports and Sanford Orthopedics and Sports Medicine. This screen includes assessments of muscle strength and movement biomechanics, along with the collection of demographic and sports participation data. Participants will then receive follow-up surveys at six and twelve months to report any new injuries.

The study is designed to provide essential normative data, which is currently lacking, particularly for tests used in the assessment of ACLR patients. This data will enhance clinicians' ability to evaluate a patient's readiness for return to sport by comparing their performance to robust normative values. Additionally, the study will collect data on other risk factors, such as a history of concussions, to better understand the interplay between these factors and biomechanics in ACL injury risk.

By establishing this comprehensive database, the study aims to improve patient care by informing ACL and ACLR treatment and return-to-play guidelines, ultimately reducing the risk of ACL re-injury in athletes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy athletes participating in formal, organized, competitive sports between the ages of 10 and 65 years old

Exclusion Criteria:

* Athletes who are injured at the time of consent and pregnant individuals

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community sampling.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2032-07-01 (Estimated); Study Completion 2033-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of injury | 6 and 12 months from baseline
  The primary outcome measure will assess the incidence of ACL injuries among participants. This metric will be determined by responses to follow-up surveys administered at 6 and 12 months post-injury risk screen. Participants will be asked whether they sustained an injury that prevented them from participating in their sport or activity for 10 or more consecutive days. The measure will capture any new ACL injuries occurring within the specified follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Bond, PhD, MBA, Principal Investigator — Sanford Health
Locations (1):
- Sanford Health, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No